CLINICAL TRIAL: NCT00115999
Title: Phase 3, Multicenter, Multi-National, Randomized, Partial Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Alfimeprase in Subjects With Acute Peripheral Arterial Occlusion
Brief Title: Study of Alfimeprase to Rapidly Dissolve Blood Clots in the Leg and Help Prevent the Need for Surgery on Leg Arteries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Brian Kersten, PhD, Nuvelo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA004; NAPA-2
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Arterial Occlusive Diseases
Keywords: PAO; acute peripheral arterial occlusion; thrombolysis; blood clot; leg attack; alfimeprase; thrombus; embolism; thromboembolism; claudication; thrombolytic; thrombosis; plasminogen activator; arterial flow
MeSH Terms: conditions — Arterial Occlusive Diseases; Thrombosis; Embolism; Thromboembolism; Intermittent Claudication | interventions — alfimeprase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alfimeprase

SUMMARY:
The purpose of this study is to directly compare the safety and efficacy of intra-thrombus alfimeprase 0.3 mg/kg with placebo in acute peripheral arterial occlusion (PAO) as measured by a 30 day open vascular free surgery rate.

DETAILED DESCRIPTION:
There is an unmet medical need to improve thrombolytic therapy in acute peripheral arterial occlusion (PAO). Currently used plasminogen activators can result in increased circulating levels of plasmin that result in a systemic "lytic state" that does not distinguish between physiologic and pathologic thrombosis. In general, mean plasminogen activator infusion durations of greater than 24 hours in order to achieve successful thrombolysis are problematic in a disease where delayed restoration of arterial flow can lead to irreversible ischemic damage. A direct thrombolytic agent like alfimeprase, with a rapid mechanism of action and a potentially safer bleeding risk profile, could facilitate a rapid restoration of arterial flow and avoidance of open vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Ages 18 or older
* Acute PAO of a lower extremity with onset of symptoms within 14 days prior to randomization
* Acute index limb ischemia classified as SVS/ISCVS Class I or IIA caused by occlusion of a native artery and/or bypass graft (vein or prosthetic)
* Need for open vascular surgical intervention in the event of unsuccessful thrombolysis
* Available for follow-up assessments

Exclusion Criteria:

* Contraindication to systemic anticoagulation
* History of endovascular procedure or open vascular surgery on the index limb within the last 30 days
* History of significant acute or chronic kidney disease that would preclude contrast angiography
* Known allergy to contrast agents
* History of heparin-induced thrombocytopenia (HIT)
* Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to randomization
* Any thrombolytic therapy within 30 days prior to randomization
* Past participation in any alfimeprase clinical trial
* History of hypersensitivity to aspirin
* Pregnant, lactating, or actively menstruating women and women of child-bearing potential who are not using adequate contraceptive precautions (e.g. intrauterine device, oral contraceptives, barrier methods, or other contraception deemed adequate by the investigator)
* Uncontrolled hypertension: systolic blood pressure (BP) > 180 mmHg, or diastolic BP > 110 mmHg at the time of baseline assessment
* Hematocrit < 30%; subjects with a low hematocrit who are not actively bleeding can be entered into this study if after transfusion their hematocrit is >= 30%
* Platelet count <100 X 10(9)/L on baseline labs
* Investigator inability to advance guidewire through index occlusion
* Medically unable to withstand an open vascular surgical procedure
* Any other feature that, in the opinion of the investigator, should preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
30 day open vascular surgery free rate

SECONDARY OUTCOMES:
Rate of arterial flow restoration at 4 hours after initiation of study drug
Rate of improvement in index limb ABI by >=0.15 at 30 days
Change in the severity of planned surgical procedures at 30 days
Change in index limb pain severity score at 30 days
30 day open vascular surgery free survival rate
Length of hospital stay
Length of intensive care unit (ICU) stay
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Deitcher, MD, Study Director — ARCA Biopharma, Inc.
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- See also: Company website — http://www.nuvelo.com